CLINICAL TRIAL: NCT06985654
Title: The Effect of Preoperative Intravenous Fluid Bolus on Post-induction Hypotension in Elective Cystoscopies.
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Principal Investigator, Sagar Bansal, Assistant Professor of Anesthesiology, University of Missouri-Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2126906
Record Dates: First submitted 2025-05-01; First posted 2025-05-22 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-05

CONDITIONS: Postinduction Hypotension; Hypotension During Surgery
Keywords: postinduction hypotension; hypotension; cystoscopy; lactated ringers
MeSH Terms: conditions — Hypotension | interventions — Ringer's Lactate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- No Treatment (No Intervention): Patients will receive an ultrasound scan on their heart to determine cardiac output before surgery, but no fluid bolus will be given.
- Preoperative Fluid Bolus (Experimental): Patients will receive an ultrasound scan on their heart to determine cardiac output and will also receive a fluid bolus of Lactated Ringers before surgery.
  Interventions: Drug: Lactated Ringers

INTERVENTIONS:
Drug: Lactated Ringers — A bolus of Lactated Ringers (15mL/kg of ideal body weight) will be given to patients prior to anesthesia induction.
  Arms: Preoperative Fluid Bolus

SUMMARY:
This study aims to determine whether a standardized, weight-based crystalloid fluid bolus administered preoperatively reduces the incidence of postinduction hypotension (PIH) in patients undergoing cystoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old.
2. Undergoing elective cystoscopy surgery as the primary procedure.
3. Able to provide informed consent.

Exclusion Criteria:

1. Emergency surgeries.
2. Past history of amputations of any body part.
3. Allergies or contraindications to any medications used in the protocol or lactated ringers.
4. Systolic heart failure with LVEF < 30% within the last year.
5. Severely depressed RV function within the last year.
6. Restrictive diastolic dysfunction within the last year.
7. Currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-07-14 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postinduction Hypotension | From the time patient enters the operating room to the end of surgery, assessed up to 24 hours.
  Number of patients that experience a decrease in mean arterial pressure (MAP) greater than 20% from the baseline MAP.

OTHER OUTCOMES:
Inferior Vena Cava Size | From the time of consent to the beginning of surgery, assessed up to 24 hours.
  Size of the inferior vena cava before surgery, approximated using a point-of-care ultrasound scan
Respiratory Variability | From the time of consent to the beginning of surgery, assessed up to 24 hours.
  Change in the size of the inferior vena cava during respiration, approximated using a point-of-care ultrasound scan

CONTACTS AND LOCATIONS:
Overall Officials: Sagar Bansal, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University Hospital, Columbia, Missouri, United States